CLINICAL TRIAL: NCT02642718
Title: Pre-operative Ketorolac Administration Has no Pre-emptive Analgesic Effect Following Total Abdominal Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Arquitecto Marcide (Other)
Responsible Party: Principal Investigator, Beatriz Nistal-Nuno, Anesthesiologist, MD, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KP 359352
Record Dates: First submitted 2015-12-19; First posted 2015-12-30 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Pain
Keywords: preemptive analgesia; postoperative pain; NSAIDs; ketorolac; abdominal hysterectomy
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): In the operating room, the anesthesiologist administered 50 mL of 0.9% saline intravenously to patients in the control group 30 minutes before surgical incision
  Interventions: Other: Placebo
- Ketorolac Tromethamine (Experimental): In the operating room, the anesthesiologist administered ketorolac (30 mg) in 50 mL of 0.9 % saline intravenously to patients in the ketorolac group 30 minutes before surgical incision. (a single dose).
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — In the operating room, the anesthesiologist administered ketorolac (30 mg) in 50 mL of 0.9 % saline intravenously to patients in the ketorolac group 30 minutes before surgical incision (a single dose).
  Other Names: ketorolac
  Arms: Ketorolac Tromethamine
Other: Placebo — In the operating room, the anesthesiologist administered 50 mL of 0.9 % saline intravenously to patients in the control group 30 minutes before surgical incision
  Arms: Placebo

SUMMARY:
Background: Experimental models using short duration noxious stimuli have led to the concept of pre-emptive analgesia. Ketorolac, a non-steroidal anti-inflammatory drug (NSAID), has been shown to have a post-operative narcotic sparing effect when given pre-operatively and alternatively to not have this effect. This study was undertaken to determine whether a single intravenous dose of ketorolac would result in decreased post-operative pain and narcotic requirements.

Methods: In a double-blind, randomized controlled trial, 48 women undergoing abdominal hysterectomy were studied. Patients in the ketorolac group received 30 mg of intravenous ketorolac 30 minutes before surgical incision, while the control group received normal saline. The post-operative analgesia was performed with a continuous infusion of tramadol at 12 mg/hour with the possibility of a 10 mg bolus every 10 minutes. Pain was assessed using the Visual Analog Scale (VAS), tramadol consumption and hemodynamic parameters at 0, 1, 2, 4, 8, 12, 16 and 24 hours post-operatively. We quantified times to rescue analgesic (morphine), adverse effects and patient satisfaction.

DETAILED DESCRIPTION:
Damage to tissues has been shown to provoke a magnified reaction to noxious stimuli, peripherally by diminishing the threshold of nociceptive afferent nerve terminals and centrally by augmenting the excitability of second-order sensory neurons in the spinal cord; later resulting in an amplification and extension of postoperative pain after surgery. Hence, much research has focused on procedures to avoid these central neuroplastic changes through the usage of preemptive analgesia.

Experimental models have conducted to the idea of 'preemptive analgesia' . The decrement of afferent nociceptive inputs to the spinal cord using analgesic techniques started before the initial painful stimulus avoids or attenuates the formation of spinal hyperexcitabilty and avoids the transformed processing of afferent input, leading to less postoperative pain. Whether such experimental models are applicable to the noxious circumstances occurring during surgery is controversial.

Although preemptive analgesia with different agents have been successful in experimental animals, conclusions from human studies remain in conflict. A diversity of agents have been analyzed for their conceivable preemptive analgesic effects: local anesthetics, non-steroidal anti-inflammatory drugs (NSAIDs), paracetamol, opioids, magnesium, cytokine synthesis inhibitors, ketamine, and tricyclic antidepressants.

Scientific research enabling an understanding of the molecular mechanisms of nociception has disclosed a considerable function of cytokines and prostaglandins (PG). Hyperexcitability also appears peripherally in nerve endings at the location of surgical tissue damage and is mediated in part by prostaglandins. Evidence is accumulating that products of the cyclooxygenase pathway may be engaged in the elaboration of central sensitization. Drugs that block the formation of prostaglandins such as NSAIDs might therefore be assumed to avoid or minimize the formation of this peripheral and central hyperexcitability. Their central analgesic actions are effected by averting spinal prostaglandin synthesis and attenuating liberation of neurotransmitters from the primary afferent terminals and spinal interneurons.

Sporadic studies have established some considerable preemptive benefit of NSAIDs. As a result, the objective of this study was to ascertain the impact of a NSAID, ketorolac, on pain severity and analgesic requirement, in the early postoperative period.

Ketorolac is a nonselective NSAID that blocks cyclooxygenase 1 (COX-1) and cyclooxygenase 2 (COX-2) enzymes and as a result blocks the formation of prostaglandins attenuating the sensitization procedures. The antinociceptive and anti-inflammatory action of NSAIDs may be associated to the suppression of nitric oxide synthase activation, decreased generation of proinflammatory cytokines, and lipoxine activation. Consequently, this multidirectional activity indicates that there may be the probability of adjusting the nociception process by the employment of these drugs perioperatively.

To our knowledge, no prior controlled study has determined the effectiveness of preoperative intravenous ketorolac compared to placebo in patients who underwent abdominal hysterectomies. Thus, this clinical trial was conceived to explore the postoperative analgesic efficiency and opioid-sparing action of a single dose of intravenous ketorolac in contrast with placebo administered preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* normal height and weight
* ASA class I, II, III
* elective surgery
* surgery time between 30-150 min
* understanding of the Visual Analog Scale (VAS)
* no allergies or intolerance to NSAIDs or anesthetics
* no psychiatric illness.

Exclusion Criteria:

* renal deterioration
* history of peptic ulceration
* asthma
* coagulopathy
* cognitive impairment
* inability to use the Patient Controlled Analgesia (PCA) device
* history of chronic pain syndromes
* history of chronic use of analgesics, sedatives, opioids or steroids
* liver or hematologic disease
* a history of drug or alcohol abuse
* therapy with NSAIDs, anticoagulants, or lithium.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-04; Primary Completion 2001-10 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Pain as measured by the Visual Analog Scale (VAS) score | at 0 hours postoperatively (arrival at recovery room)
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Pain as measured by the Visual Analog Scale (VAS) score | at 1 hour postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Pain as measured by the Visual Analog Scale (VAS) score | at 2 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Pain as measured by the Visual Analog Scale (VAS) score | at 4 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Pain as measured by the Visual Analog Scale (VAS) score | at 8 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Pain as measured by the Visual Analog Scale (VAS) score | at 12 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Pain as measured by the Visual Analog Scale (VAS) score | at 16 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Pain as measured by the Visual Analog Scale (VAS) score | at 24 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).

SECONDARY OUTCOMES:
tramadol consumption | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  The cumulative amounts of tramadol (mg) administered through the Patient-Controlled-Analgesia (PCA) device as a basal infusion and the incremental supplemental bolus required by the patient were documented at these time points.

OTHER OUTCOMES:
Blood Pressure (BP) systolic | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  Measured in mm Hg. We evaluated these hemodynamic parameters as an indirect measure of pain.
Blood Pressure (BP) diastolic | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  Measured in mm Hg. We evaluated these hemodynamic parameters as an indirect measure of pain
Heart rate | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  We evaluated these hemodynamic parameters as an indirect measure of pain
Respiratory rate | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  We evaluated these hemodynamic parameters as an indirect measure of pain.
Time for the first demand of analgesia | 24 h postoperatively.
  The time interval to first solicited rescue analgesia in the 24 h postoperatively (in minutes). This rescue analgesia was administered if the established analgesic treatment was not sufficient to alleviate pain.
Number of rescue doses | 24 h postoperatively
  The number of times a rescue analgesic dose was administered as a supplement in the first postoperative 24 hours.
Satisfaction score | 24 hours postoperatively
  Global patient satisfaction (0-3), regarding pain control, was measured 24 hours after the operation
Side effects | 24 hours postoperatively
  Number of Participants with Serious and Non-Serious Adverse Events in the 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Nistal-Nuño, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (2):
- Complexo Hospitalario Arquitecto Marcide-Prof. Novoa Santos, Ferrol, A Coruña, Spain
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No